CLINICAL TRIAL: NCT04096027
Title: Cabergoline Before or After Oocyte Collection for Follicular Resolution
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fertility Center of Las Vegas (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19-FCLV-101
Record Dates: First submitted 2019-09-16; First posted 2019-09-19 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — Cabergoline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Laboratory personnel will not be informed of the subject's group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early administration (Experimental): Cabergoline administered the day before egg collection.
  Interventions: Drug: Cabergoline Pill
- Late administration (Experimental): Cabergoline administered after egg collection.
  Interventions: Drug: Cabergoline Pill

INTERVENTIONS:
Drug: Cabergoline Pill — 0.5 mg cabergoline pill taken orally

SUMMARY:
Randomized trial comparing the efficacy of two different times of administration of cabergoline in patients undergoing controlled ovarian stimulation and oocyte collection.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female at least 18 years of age intending to undergo ovarian stimulation for a cycle of IVF.
2. Ability read and understand English sufficiently to obtain informed consent and complete a study diary.
3. Pre-implantation genetic screening (PGS) is allowed.
4. Egg donors are allowed.
5. Patients using a gestational carrier are allowed.
6. Patients with prior IVF cycles are allowed, but no patient can undergo more than one cycle with oocyte collection under this study.

Exclusion Criteria:

1. Egg banking, donor egg banking, or any cycle type that would preclude immediate culture to blastocyst stage.
2. Patients that would be unavailable for the follow-up ultrasound 5 days post-retrieval, such as patients that live far from the clinic (e.g. out of state).
3. Uncontrolled hypertension.
4. Ergot alkaloid hypersensitivity or allergy.
5. History of pulmonary, pericardial, retroperitoneal fibrotic disorders.
6. History of bipolar disorder, schizophrenia, or psychotic illness.
7. Breast feeding.
8. History of eclampsia or pre-eclampsia.
9. Severe hepatic dysfunction.
10. Current use of any dopamine receptor agonist or antagonist for any purpose, including, but not limited to, cabergoline (Dostinex), aripiprazole (Abilify), bromocriptine (Parlodel), methylphenidate (Ritalin), buproprion (Wellbutrin, Zyban), lisdexamfetamine (Vyvanse).
11. Any condition that, in the opinion of the physician or principal investigator, would place the patient at undue risk under this protocol or would otherwise make the protocol inappropriate for that subject.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

PRIMARY OUTCOMES:
Discomfort level | 5 days after egg collection
  Self-assessed discomfort level
Mature oocyte rate per follicular puncture | Within 24 hours of egg collection
  Ratio of mature oocytes obtained to punctured ovarian follicles

SECONDARY OUTCOMES:
Ovarian volume | 5 days post retrieval
oocyte count | Within 24 hours of egg collection
Oocyte to follicle ratio | Within 24 hours of egg collection
M1 oocyte rate | Within 24 hours of egg collection
M1 to M2 oocyte ratio | Within 24 hours of egg collection
Aneuploidy rate | Within 14 days of egg collection
  Genetic test results of embryos for patients who opt for such testing.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Shapiro, MD, Principal Investigator — Fertility Center of Las Vehas
Locations (1):
- Fertility Center of Las vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No